CLINICAL TRIAL: NCT05851391
Title: buRst-supprESsion TO Stop Refractory Status Epilepticus Post-cardiac Arrest (RESTORE)
Brief Title: buRst-supprESsion TO Stop Refractory Status Epilepticus Post-cardiac Arrest
Acronym: RESTORE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The ZOLL Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-34336
Record Dates: First submitted 2023-02-24; First posted 2023-05-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypoxia-Ischemia, Brain; Heart Arrest; Status Epilepticus; Refractory Status Epilepticus; Seizures; Anoxic-Ischemic Encephalopathy; Anoxia-Ischemia, Cerebral
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest; Status Epilepticus; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Burst Suppression EEG Target (Other): Anesthetic will be titrated to achieve burst suppression on continuous EEG (50-99% attenuation/suppression) for 24 hours.
  Interventions: Drug: Burst Suppression EEG Target Intravenous Anesthesia
- Seizure Suppression EEG Target (Other): Anesthetic will be titrated to achieve seizure suppression on continuous EEG for 24 hours.
  Interventions: Drug: Seizure Suppression EEG Target Intravenous Anesthesia

INTERVENTIONS:
Drug: Burst Suppression EEG Target Intravenous Anesthesia — The objective of the burst suppression EEG target is to stop seizures by titrating the anesthetic infusion to suppress most of the EEG background (>50% suppressed/attenuated). After this 24-hour period, this target would be continued for 24 hours. The anesthetic will then be tapered under EEG monitoring. In case of PCARSE recurrence, the intervention with the same target will be re-initiated for another cycle of 24 hours.
  Arms: Burst Suppression EEG Target
Drug: Seizure Suppression EEG Target Intravenous Anesthesia — is to stop seizures by titrating the anesthetic infusion without suppressing most of the EEG background. This target would be continued for 24 hours. After this 24-hours period, this target would be continued for 24 hours. The anesthetic will then be tapered under EEG monitoring. In case of PCARSE recurrence, the intervention with the same target will be re-initiated for another cycle of 24 hours.
  Arms: Seizure Suppression EEG Target

SUMMARY:
RESTORE is a randomized clinical trial investigating the safety and feasibility of using EEG treatment targets (burst suppression vs. seizure suppression) for post-cardiac arrest refractory status epilepticus treatment.

DETAILED DESCRIPTION:
Rationale: Seizures emerge as a complication of hypoxic-ischemic brain injury in near a third of patients successfully resuscitated from cardiac arrest. Seizures post-cardiac arrest can be refractory to treatment with anti-seizure medications and anesthetics may be used for refractory status epilepticus control. Anesthetic treatment guided by continuous EEG can target burst suppression or seizure suppression, however it is not known which strategy is superior for achieving PCARSE control.

Objective: determine the safety and feasibility of post-cardiac arrest refractory status epilepticus (PCARSE) treatment using EEG goals for intravenous anesthetic titration (burst suppression vs. seizure suppression).

Clinical Trial Phase: II

Study Design: prospective, randomized, open-label, blinded end-point, concurrently-controlled, parallel arms design clinical trial.

Study Period: two years

Study Population: unconscious cardiac arrest survivors with return of spontaneous circulation who develop post-cardiac arrest refractory status epilepticus (PCARSE).

Interventions: anesthetic use targeting burst suppression vs. seizure suppression on EEG for 24 hours. Intervention maybe repeated using the dame EEG target once in case of PCARSE recurrence.

Sample Size: 30 subjects randomized in a 1:1 ratio to either burst suppression or seizure suppression EEG targets.

Primary Endpoints: Safety and feasibility of seizure control using burst suppression or seizure suppression EEG targets for PCARSE treatment.

Secondary Endpoints: Seizure recurrence incidence, time to seizure recurrence, number and dose of anti-seizure medication and anesthetic needed for PCARSE control, Death or disability according to the Cerebral Performance Category at Discharge (30 days), and Death or disability according to the modified Rankin Scale at Discharge (30 days).

Risks: Participants receiving anesthetics for PCARSE treatment will be monitored for hypotension, propofol infusion syndrome, and hypertriglyceridemia. Patients with PCARSE are at high risk for death and prolonged hospital stays.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Non-traumatic, out-of-hospital cardiac arrest
3. Comatose on admission - defined as not following commands
4. Return of spontaneous circulation (ROSC) within less than 45 minutes
5. Admission to the intensive care unit
6. Diagnosis of post-cardiac arrest refractory status epilepticus confirmed with continuous

EEG monitoring within 7 days from ROSC

Exclusion Criteria:

1. Acute cerebral hemorrhage or infarction
2. Pregnancy
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-cardiac arrest refractory status epilepticus control | 48 hours
  Continuous EEG will be monitored to determine time to PCARSE recurrence during the anesthetic maintenance and anesthetic weaning phase (combined)

SECONDARY OUTCOMES:
Seizure recurrence incidence and duration (burden) | 24-48 hours
  Presence of seizures on EEG after initiation of anesthetic maintenance phase
Neurological Function at Discharge (CPC: Cerebral Performance Category) | 30 days
  Cerebral Performance Category score at Discharge
Neurological Function at Discharge (mRS: modified Ranking Scale) | 30 days
  modified Rankin Scale score at Discharge
Neurological Function 90 days (CPC: Cerebral Performance Category) | 90 days
  Cerebral Performance Category score at 90 days
Neurological Function 90 days (mRS: modified Ranking Scale) | 90 days
  modified Rankin Scale score at Discharge
Neurological Function 180 days (mRS: modified Ranking Scale) | 180 days
  modified Rankin Scale score at Discharge
Neurological Function180 days (mRS: modified Ranking Scale) | 180 days
  modified Rankin Scale score at Discharge
PCARSE Treatment Intensity | 24-48 hours
  Number of anti-seizure medications and anesthetics used for PCARSE control after initiation of anesthetic maintenance phase and prior to weaning
Seizure recurrence incidence and duration (burden) | 24-48 hours
  Presence of seizures on EEG after initiation of anesthetic weaning phase
PCARSE Treatment Intensity | 24-48 hours
  Dose of anti-seizure medications and anesthetics used for PCARSE control after initiation of anesthetic maintenance phase and prior to weaning

CONTACTS AND LOCATIONS:
Overall Officials: Edilberto Amorim, MD, Principal Investigator — Assistant Professor of Neurology
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No